CLINICAL TRIAL: NCT05884840
Title: Health Program for prEvention of cardiovascuLar disEases Based on a Risk screeNing Strategy With Ankle-brachial Index.
Brief Title: New Cardiovascular Risk Screening Strategy.
Acronym: HELENA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Hospital del Mar Research Institute (IMIM) (Other); Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other); Institut Català de la Salut (Other); Biobizkaia Health Research Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SLT/21/000015
Record Dates: First submitted 2023-05-10; First posted 2023-06-01 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Cardiovascular Prevention; Screening; Peripheral Artery Disease; Arteriosclerosis; Asymptomatic
MeSH Terms: conditions — Peripheral Arterial Disease; Arteriosclerosis

STUDY DESIGN:
Intervention Model Description: This study will be conducted as a clustered randomized pragmatic clinical trial (CRT) in primary care practice. During the period of two years (2023-2025), randomization of the eight Health Regions (274 primary care centres) in Catalonia will take place. The current strategy, in Catalonia, for cardiovascular risk screening is based on risk assessment using Framingham-REGICOR risk function. In the intervention group, a screening program with ABI will be added to all 50-74-year-old individuals with Framingham-REGICOR risk ≥7% and high probability of having ABI≤0.9. The probability of having ABI≤0.9 will be estimated using the REASON function and will be defined as a probability ≥7%. People that are classified as ABI≤0.9 high-risk, will undergo a PAD screening program using ABI test. If the result of the ABI is equal and lower than 0.9, indications of the Health Catalan Institute's CV and lipid guidelines will be recommended by physicians to the patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group PAD screening program (Experimental): Patients aged 50-74 years free of any symptomatic or history of CVD and a Framingham-REGICOR risk ≥7%, will be candidates for PAD screening program using REASON's function predicative capacity
  Interventions: Diagnostic Test: HELENA
- Control group PAD screening program (No Intervention): Patients aged 50-74 years free of any symptomatic or history of CVD will be candidates as a comparison group to calculate the cost-utility and reduction of CVD risk and events.

INTERVENTIONS:
Diagnostic Test: HELENA — The current CV risk screening program in based using the REGICOR risk function, which is integrated in the primary care electronic health record. This risk function predicts the probability within 10 years of developing a coronary event. Those who are categorized as high risk, obtaining a 10% of probability, are candidates of receiving lipid lowering drugs and recommendations on healthy life habits.
  What this intervention suggests is that, besides the REGICOR estimation, the electronic health records will also incorporate a new CV risk function, REASON. The model predicts the risk of holding a pathologic ABI score, in people aged 50-74 years old who are apparently free of CV. Patients who obtain a score ≥ 7 will undergo a PAD screening program with ABI test. If the value of the test is ≤0.9, the REGICOR, physicians will recommend indications of the Health Catalan Institute's CV and lipid Guidelines to the patients.
  Arms: Intervention group PAD screening program

SUMMARY:
Mortality due to cardiovascular disease (CVD) in Spain accounted for 29% of all deaths (32% in women and 26% in men) in 2017. Out of those, 67% were related to a coronary or a cerebrovascular disease .

A key strategy in primary prevention of CVD is to use risk functions to individualize preventive interventions for each patient. The current CV risk-screening program in some regions of Spain, is based using an adapted Framingham scale, REGICOR's risk function, which is integrated in the primary care electronic health record. This risk function predicts the probability within 10 years of developing a coronary event. However, this function fails to identify patients that fall into low- or intermediate-risk level, and might develop a CV event in the up following 10 years.

Ankle-brachial index (ABI) is a simple, non-invasive and economic technique, which allows detecting peripheral arterial disease (PAD), and gives independent risk function information compared to other coronary risk functions. Even tough, between 13-27% of middle age population have an ABI ≤ 9, around 50-89% of them do not exhibit any symptoms. However, they hold higher mortality risk and CV events. Current clinical guidelines for PAD screening, have a limited level of evidence, and only recommend using ABI on patients aged 50-70, who have diabetes or are smokers, and patients older than 70 years old.

A new risk function, REASON, to assess CVD risk has been designed. This model has proven to improve predictive capacity of holding an ABI ≤ 0.9 on those patients aged 50-74 that are apparently free of CVD. Therefore, a strategy that combines the current CV risk estimation using REGICOR, and the prediction capacity of pathologic ABI with REASON, would allow detecting high-risk patients with a PAD screening program. It is possible that patients, who hold an ABI ≤ 0.9, even if being asymptomatic, will adopt physician's recommendations on healthy life habits and preventive treatment.

The aims of this study are:

* To assess the effectiveness and cost-utility of adding a screening program with ABI to the current strategy of CV risk detection to reduce the incidence of CVD and mortality from all causes in the population aged 50 to 74.
* To assess the effectiveness of adding a screening program with ABI to the current strategy of CV risk detection to improve cardiovascular risk factors in the population aged 50 to 74.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50 to 74, which are free or do not have previous history of CVD. Patients that hold a REGICOR CV risk score ≥7, and REASON risk core ≥7, during a routine primary care visit

Exclusion Criteria:

* Symptomatic PAD
* Coronary disease
* Stroke
* Cardiac revascularization

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54000 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Hard coronary heart disease (CHD) | 3 years
  Myocardial infarction, cardiac revascularization, or coronary death
Major adverse cardiovascular event (MACE) | 3 years
  A composite of hard CHD (myocardial infarction, cardiac revascularization, or coronary death) and stroke (fatal and nonfatal ischemic stroke)
All-cause mortality | 3 years
Tabaco consumption (CVD risk factors improvement assessment) | 3 years
  Smoker, ex-smoker or non-smoker
Lipid profile (CVD risk factors improvement assessment) | 3 years
  Total cholesterol (mg/dl), LDL (mg/dl), HDL (mg/dl), Triglycerides (mg/dl)
Systolic and diastolic pressure (CVD risk factors improvement assessment) | 3 years
  mm Hg
Weight (CVD risk factors improvement assessment) | 3 years
  kg
Height (CVD risk factors improvement assessment) | 3 years
  m
BMI (CVD risk factors improvement assessment) | 3 years
  (kg/m2) Will be calculated dividing the weight in kilograms by their height in metres squared
Glycaemia (CVD risk factors improvement assessment) | 3 years
  Fasting blood sugar (mg/dl)
Glycated haemoglobin (CVD risk factors improvement assessment) | 3 years
  (in DM patients) glycosylated hemoglobin in the blood (mg/dl) or percentage (%)
Creatinine (CVD risk factors improvement assessment) | 3 years
  mg/dL
Proteinuria (CVD risk factors improvement assessment) | 3 years
  mg/dL protein in urine
Albumin-to-creatinine ratio (ACR) (CVD risk factors improvement assessment) | 3 years
  ACR (mg/g) will be calculated by by dividing mg of proteinuria (albumine) by g of creatinine.
Glomerular filtrate rate (CVD risk factors improvement assessment) | 3 years
  Levels of creatinine in milliliters of cleansed blood per minute per body surface (mL/min/1.73m2).

SECONDARY OUTCOMES:
Coronary heart disease | 3 years
  A composite of angina and hard CHD
Cerebrovascular disease | 3 years
  A composite of stroke (fatal and nonfatal ischemic stroke) and transient ischemic attack
Cardiovascular disease | 3 years
  a composite of MACE, angina and transient ischemic attack
Lipid lowering medication Adverse effects | 3 years
  1) Short-term effects: Muscular and hepatic alterations, and 2) long-term effects: Diabetes and cancer

CONTACTS AND LOCATIONS:
Overall Officials: Rafel Ramos Blanes, MD, PhD, Principal Investigator — Unidad de Investigación en Atención Primaria de Girona, IDIAP Jordi Gol
Locations (1):
- Institut Català de la Salut (ICS), Barcelona, Spain

REFERENCES:
- [Background] Ministerio de Sanidad SS e I. Indicadores de Salud 2020 Evolución de los indicadores del estado de salud en España y su magnitud en el contexto de la Unión Europea. Madrid; 2020.
- [Background] Institute for Health Metrics and Evaluation. Global Burden of Disease Results Tool, Global Health Data Exchange. 2017
- [Background] Wilkins E, et al. European Cardiovascular Disease Statistics. European Heart Network, editor. Brussels; 2017
- [Background] Visseren FLJ, Mach F, Smulders YM, Carballo D, Koskinas KC, Back M, Benetos A, Biffi A, Boavida JM, Capodanno D, Cosyns B, Crawford C, Davos CH, Desormais I, Di Angelantonio E, Franco OH, Halvorsen S, Hobbs FDR, Hollander M, Jankowska EA, Michal M, Sacco S, Sattar N, Tokgozoglu L, Tonstad S, Tsioufis KP, van Dis I, van Gelder IC, Wanner C, Williams B; ESC National Cardiac Societies; ESC Scientific Document Group. 2021 ESC Guidelines on cardiovascular disease prevention in clinical practice. Eur Heart J. 2021 Sep 7;42(34):3227-3337. doi: 10.1093/eurheartj/ehab484. No abstract available. PMID 34458905
- [Background] Comin E, Solanas P, Cabezas C, Subirana I, Ramos R, Gene-Badia J, Cordon F, Grau M, Cabre-Vila JJ, Marrugat J. [Estimating cardiovascular risk in Spain using different algorithms]. Rev Esp Cardiol. 2007 Jul;60(7):693-702. Spanish. PMID 17663853
- [Background] Morrow DA, de Lemos JA. Benchmarks for the assessment of novel cardiovascular biomarkers. Circulation. 2007 Feb 27;115(8):949-52. doi: 10.1161/CIRCULATIONAHA.106.683110. No abstract available. PMID 17325253
- [Background] Grewal J, Anand S, Islam S, Lonn E; SHARE and SHARE-AP Investigators. Prevalence and predictors of subclinical atherosclerosis among asymptomatic "low risk" individuals in a multiethnic population. Atherosclerosis. 2008 Mar;197(1):435-42. doi: 10.1016/j.atherosclerosis.2007.06.020. Epub 2007 Aug 6. PMID 17675040
- [Background] Greenland P, Abrams J, Aurigemma GP, Bond MG, Clark LT, Criqui MH, Crouse JR 3rd, Friedman L, Fuster V, Herrington DM, Kuller LH, Ridker PM, Roberts WC, Stanford W, Stone N, Swan HJ, Taubert KA, Wexler L. Prevention Conference V: Beyond secondary prevention: identifying the high-risk patient for primary prevention: noninvasive tests of atherosclerotic burden: Writing Group III. Circulation. 2000 Jan 4;101(1):E16-22. doi: 10.1161/01.cir.101.1.e16. No abstract available. PMID 10618318
- [Background] McDermott MM, Greenland P, Liu K, Guralnik JM, Celic L, Criqui MH, Chan C, Martin GJ, Schneider J, Pearce WH, Taylor LM, Clark E. The ankle brachial index is associated with leg function and physical activity: the Walking and Leg Circulation Study. Ann Intern Med. 2002 Jun 18;136(12):873-83. doi: 10.7326/0003-4819-136-12-200206180-00008. PMID 12069561
- [Background] Ramos R, Quesada M, Solanas P, Subirana I, Sala J, Vila J, Masia R, Cerezo C, Elosua R, Grau M, Cordon F, Juvinya D, Fito M, Isabel Covas M, Clara A, Angel Munoz M, Marrugat J; REGICOR Investigators. Prevalence of symptomatic and asymptomatic peripheral arterial disease and the value of the ankle-brachial index to stratify cardiovascular risk. Eur J Vasc Endovasc Surg. 2009 Sep;38(3):305-11. doi: 10.1016/j.ejvs.2009.04.013. Epub 2009 Jun 10. PMID 19515589
- [Background] Heald CL, Fowkes FG, Murray GD, Price JF; Ankle Brachial Index Collaboration. Risk of mortality and cardiovascular disease associated with the ankle-brachial index: Systematic review. Atherosclerosis. 2006 Nov;189(1):61-9. doi: 10.1016/j.atherosclerosis.2006.03.011. Epub 2006 Apr 18. PMID 16620828
- [Background] Ankle Brachial Index Collaboration; Fowkes FG, Murray GD, Butcher I, Heald CL, Lee RJ, Chambless LE, Folsom AR, Hirsch AT, Dramaix M, deBacker G, Wautrecht JC, Kornitzer M, Newman AB, Cushman M, Sutton-Tyrrell K, Fowkes FG, Lee AJ, Price JF, d'Agostino RB, Murabito JM, Norman PE, Jamrozik K, Curb JD, Masaki KH, Rodriguez BL, Dekker JM, Bouter LM, Heine RJ, Nijpels G, Stehouwer CD, Ferrucci L, McDermott MM, Stoffers HE, Hooi JD, Knottnerus JA, Ogren M, Hedblad B, Witteman JC, Breteler MM, Hunink MG, Hofman A, Criqui MH, Langer RD, Fronek A, Hiatt WR, Hamman R, Resnick HE, Guralnik J, McDermott MM. Ankle brachial index combined with Framingham Risk Score to predict cardiovascular events and mortality: a meta-analysis. JAMA. 2008 Jul 9;300(2):197-208. doi: 10.1001/jama.300.2.197. PMID 18612117
- [Background] Espinola-Klein C, Rupprecht HJ, Bickel C, Lackner K, Savvidis S, Messow CM, Munzel T, Blankenberg S; AtheroGene Investigators. Different calculations of ankle-brachial index and their impact on cardiovascular risk prediction. Circulation. 2008 Aug 26;118(9):961-7. doi: 10.1161/CIRCULATIONAHA.107.763227. Epub 2008 Aug 12. PMID 18697822
- [Background] US Preventive Services Task Force; Curry SJ, Krist AH, Owens DK, Barry MJ, Caughey AB, Davidson KW, Doubeni CA, Epling JW Jr, Kemper AR, Kubik M, Landefeld CS, Mangione CM, Silverstein M, Simon MA, Tseng CW, Wong JB. Screening for Peripheral Artery Disease and Cardiovascular Disease Risk Assessment With the Ankle-Brachial Index: US Preventive Services Task Force Recommendation Statement. JAMA. 2018 Jul 10;320(2):177-183. doi: 10.1001/jama.2018.8357. PMID 29998344
- [Background] Norgren L, Hiatt WR, Dormandy JA, Nehler MR, Harris KA, Fowkes FG; TASC II Working Group; Bell K, Caporusso J, Durand-Zaleski I, Komori K, Lammer J, Liapis C, Novo S, Razavi M, Robbs J, Schaper N, Shigematsu H, Sapoval M, White C, White J, Clement D, Creager M, Jaff M, Mohler E 3rd, Rutherford RB, Sheehan P, Sillesen H, Rosenfield K. Inter-Society Consensus for the Management of Peripheral Arterial Disease (TASC II). Eur J Vasc Endovasc Surg. 2007;33 Suppl 1:S1-75. doi: 10.1016/j.ejvs.2006.09.024. Epub 2006 Nov 29. No abstract available. PMID 17140820
- [Background] Ramos R, Baena-Diez JM, Quesada M, Solanas P, Subirana I, Sala J, Alzamora M, Fores R, Masia R, Elosua R, Grau M, Cordon F, Pera G, Rigo F, Marti R, Ponjoan A, Cerezo C, Brugada R, Marrugat J. Derivation and validation of REASON: a risk score identifying candidates to screen for peripheral arterial disease using ankle brachial index. Atherosclerosis. 2011 Feb;214(2):474-9. doi: 10.1016/j.atherosclerosis.2010.11.015. Epub 2010 Nov 19. PMID 21167488
- [Background] Perlstein TS, Creager MA. The ankle-brachial index as a biomarker of cardiovascular risk: it's not just about the legs. Circulation. 2009 Nov 24;120(21):2033-5. doi: 10.1161/CIRCULATIONAHA.109.907238. Epub 2009 Nov 9. No abstract available. PMID 19901185
- [Background] Ramos R, Garcia-Gil M, Comas-Cufi M, Quesada M, Marrugat J, Elosua R, Sala J, Grau M, Marti R, Ponjoan A, Alves-Cabratosa L, Blanch J, Bolibar B. Statins for Prevention of Cardiovascular Events in a Low-Risk Population With Low Ankle Brachial Index. J Am Coll Cardiol. 2016 Feb 16;67(6):630-640. doi: 10.1016/j.jacc.2015.11.052. PMID 26868687
- [Background] Lindholt JS, Sogaard R. Population screening and intervention for vascular disease in Danish men (VIVA): a randomised controlled trial. Lancet. 2017 Nov 18;390(10109):2256-2265. doi: 10.1016/S0140-6736(17)32250-X. Epub 2017 Aug 28. PMID 28859943
- [Background] Diederichsen AC, Rasmussen LM, Sogaard R, Lambrechtsen J, Steffensen FH, Frost L, Egstrup K, Urbonaviciene G, Busk M, Olsen MH, Mickley H, Hallas J, Lindholt JS. The Danish Cardiovascular Screening Trial (DANCAVAS): study protocol for a randomized controlled trial. Trials. 2015 Dec 5;16:554. doi: 10.1186/s13063-015-1082-6. PMID 26637993
- [Background] Betriu A, Farras C, Abajo M, Martinez-Alonso M, Arroyo D, Barbe F, Buti M, Lecube A, Portero M, Purroy F, Torres G, Valdivielso JM, Fernandez E. Randomised intervention study to assess the prevalence of subclinical vascular disease and hidden kidney disease and its impact on morbidity and mortality: The ILERVAS project. Nefrologia. 2016 Jul-Aug;36(4):389-96. doi: 10.1016/j.nefro.2016.02.008. Epub 2016 Apr 1. English, Spanish. PMID 27044887
- [Derived] Dominguez-Armengol G, Ribas-Aulinas F, Ballo E, Alzamora-Sas M, Serrat-Costa M, Ruiz-Comellas A, Forcadell-Peris MJ, Toran P, Marti-Lluch R, Ponjoan A, Blanch J, Alves-Cabratosa L, Zacarias-Pons L, Tornabell-Noguera E, Sanchez-Perez A, Berenguera-Osso A, Ramos R; HELENA Study Group. Health program for prEvention of cardiovascuLar disEases based on a risk screeNing strategy with Ankle-brachial index: HELENA study protocol. Front Public Health. 2025 May 30;13:1484163. doi: 10.3389/fpubh.2025.1484163. eCollection 2025. PMID 40520295